CLINICAL TRIAL: NCT03434665
Title: Transradial Selective Catheterization of the Celiac Artery in Obese Patients: A Pilot Study
Brief Title: Transradial Selective Catheterization of the Celiac Artery in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Olivier F. Bertrand, MD PhD; Interventional Cardiologist, Quebec Heart-Lung Institute; Associate-Professor, Faculty of Medicine, Laval University, Laval University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EASY-AngioBar
Record Dates: First submitted 2018-01-30; First posted 2018-02-15 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Obesity
Keywords: Angiography; Bariatric embolization; Gastric artery; Obesity; Transradial
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Feasibility pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recruited patients (Other): Transradial celiac artery angiography
  Interventions: Procedure: Transradial celiac artery angiography

INTERVENTIONS:
Procedure: Transradial celiac artery angiography — * After completion of transradial diagnostic coronary angiography and/or PCI, before removal of the radial arterial sheath, selective angiography of the celiac artery will be performed.
  * Technically, a 0.35-inch wire is advanced into the descending aorta. A 125 cm 5-French Judkins right catheter is inserted over this wire, which is then removed. The distal tip of the catheter is brought in front of the ostium of the celiac artery and positioning is confirmed with angiography of the celiac artery. Two or three views will be obtained to determine the optimal view to visualize the left gastric artery anatomy. All material is removed and hemostasis is obtained as per clinical routine for coronary angiography.

SUMMARY:
BACKGROUND:

* Obesity, with its associated comorbidities, is set to become a major risk factor for cardiovascular disease in the 21st century. To this day, diet and medical therapy have proven only limited efficacy and bariatric surgery remains the last resort for many severely obese patients who wish to lose weight, modify their cardiovascular risk factors and ultimately modify their long-term prognosis. However, bariatric surgery remains associated with significant procedural morbidity and many patients are not eligible for such a surgery procedure as the risk-benefit ratio of bariatric surgery in severe obese patients with coronary artery disease is not yet well known.
* Recently, percutaneous left gastric artery embolization has been reported as a promising technique leading to a body weight loss that is equivalent to bariatric surgery.
* In the context of an endovascular procedure in obese patients, vascular access is a major concern. Transradial access (or radial artery approach) has been consistently associated with significant reductions in access-site related vascular complications and peri-procedural bleeding compared to the standard transfemoral access (or femoral artery approach). This is particularly evident in patients with severe obesity.
* Visceral arteries most often have an acute angulation with the aorta which makes them more easily cannulated from above (transradial access) compared to below (transfemoral access). Preliminary experience has shown that cannulation of the celiac artery is feasible from transfemoral and transradial access, the latter being associated with shorter procedural time and less contrast agent use. To date, several pilot studies have reported successful percutaneous embolization of the left gastric artery with biodegradable microspheres. This appears to be a promising technique to reduce weight in severely obese patients.
* Prior to launching a randomized trial, further study is warranted regarding the feasibility and safety aspects of transradial angiography of the celiac artery.

DETAILED DESCRIPTION:
RATIONALE:

* A significant proportion of patients referred to IUCPQ-UL catheterization laboratory are overweight (body mass index >25 kg/m²).
* Ongoing research and early clinical experience suggest that embolization of the left gastric artery could drastically reduce ghrelin levels and be associated with significant weight loss.
* In obese patients, catheterization using femoral artery access is associated with higher risks of vascular complications and peri-procedural bleeding compared to a radial artery approach.
* Given the anatomy (angle) of the celiac artery, selective catheterization of the celiac and left gastric arteries remains challenging, especially in obese patients.
* Before studying the effects of bariatric embolization, more data regarding the access of the left gastric artery is necessary.

HYPOTHESES:

* Transradial angiography of the celiac artery/left gastric artery is feasible and safe.
* Given the angulation of celiac artery, catheterization through a radial approach could be simpler.
* Selective angiography of the celiac artery and the left gastric artery can be performed in the setting of uncomplicated coronary angiography/percutaneous coronary intervention (PCI).
* Detailed anatomy of the celiac artery and its branches can be visualized by selective transradial angiography.

OBJECTIVES:

* The primary objective is to demonstrate the feasibility and safety of performing selective angiography of the celiac artery using a transradial approach in obese patients referred for diagnostic coronary angiography and/or PCI.
* The secondary objective is to observe anatomical variations of the celiac artery and the left gastric artery.

STUDY DESIGN:

> A prospective pilot study performed at Quebec Heart & Lung Institute (Institut Universitaire de Cardiologie et de Pneumologie de Québec - Université Laval; IUCPQ-UL).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing coronary angiography with a BMI >30 kg/m² will be eligible.

Exclusion Criteria:

* Kidney disease defined by a glomerular filtration rate less than 60 ml/min/m² according to the Modification of Diet in Renal Disease (MDRD) formula;
* Previous gastric or bariatric surgery;
* Emergency coronary procedure.

Furthermore, the procedure will be cancelled if one of the following criteria are met during the coronary angiography:

* Contrast volume >250 ml;
* Radiation dose >180 Gy.cm² as assessed by the dose area product (DAP).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-02-09 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Percentage of successful selective angiographies | Baseline
  The primary end-point will be the percentage of successful selective angiographies of the celiac artery.

SECONDARY OUTCOMES:
Incidence of complications of angiographies | Baseline
  As catheterization and angiography of the celiac artery is an endovascular procedure, the incidence of vessel trauma (such as dissection or perforation) during the procedure will be assessed. All cine films will be reviewed by a multidisciplinary team.
Procedure duration | Baseline
  Time (minutes) required to complete the angiography of the celiac artery
Contrast volume | Baseline
  Volume (mL) of contrast required to complete the angiography of the celiac artery
Radiation exposure (duration) | Baseline
  Fluoroscopy time (minutes) required to complete the angiography of the celiac artery
Radiation exposure (dose) | Baseline
  Dose area product (Gy·cm2) required to complete the angiography of the celiac artery
Number of catheters | Baseline
  The number of catheters required to complete the angiography of the celiac artery

CONTACTS AND LOCATIONS:
Overall Officials: Olivier F Bertrand, MD PhD, Principal Investigator — IUCPQ-UL and Laval University
Locations (1):
- Quebec Heart & Lung Institute (IUCPQ-UL), Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided
To be completed